CLINICAL TRIAL: NCT02218515
Title: Evaluation of Gingival Crevicular Fluid Transforming Growth Factor-β1 Level After Treatment of Intrabony Periodontal Defects With Enamel Matrix Derivatives and Autogenous Bone Graft
Brief Title: Treatment of Intrabony Periodontal Defects With Enamel Matrix Derivatives and Autogenous Bone Graft
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haner Direskeneli, Prof (Other)
Responsible Party: Sponsor-Investigator, Haner Direskeneli, Prof, Prof. Dr., Marmara University
Organization: Marmara University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAG-C-DRP-090909-0288
Record Dates: First submitted 2014-08-11; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Periodontal Bone Loss; Chronic Periodontitis
Keywords: Autogenous bone graft; Chronic periodontitis; Enamel matrix derivatives; Gingival crevicular fluid; Periodontal flap surgery
MeSH Terms: conditions — Alveolar Bone Loss; Chronic Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Open Flap Debridement (Other): Open Flap Debridement (Control Group)
  Interventions: Procedure: Open Flap Debridement
- Enamel Matrix Derivative (Experimental): Open Flap Debridement+EmdogainⓇ(Enamel Matrix Derivative)
  Interventions: Biological: EmdogainⓇ(Enamel Matrix Derivative)
- Enamel Matrix Derivative+Autogenous Bone (Experimental): Open Flap Debridement+EmdogainⓇ(Enamel Matrix Derivative)+Autogenous Bone
  Interventions: Biological: EmdogainⓇEnamel Matrix Derivative+Autogenous Bone

INTERVENTIONS:
Procedure: Open Flap Debridement — Open Flap Debridement (Control Group)
  Arms: Open Flap Debridement
Biological: EmdogainⓇ(Enamel Matrix Derivative) — Open Flap Debridement+Enamel Matrix Derivative
  Arms: Enamel Matrix Derivative
Biological: EmdogainⓇEnamel Matrix Derivative+Autogenous Bone — Open Flap Debridement+EmdogainⓇ(Enamel Matrix Derivative)+Autogenous Bone
  Arms: Enamel Matrix Derivative+Autogenous Bone

SUMMARY:
The present study aimed to evaluate the effects of enamel matrix derivatives either alone or combined with autogenous bone graft applied to intrabony defects in chronic periodontitis patients on clinical/radiographic parameters and gingival crevicular fluid transforming growth factor-β1 level and, to compare with open flap debridement. Our hypothesis is to test whether the use of autogenous bone graft and enamel matrix derivative combination in the treatment of intrabony periodontal defects enhance the clinical, radiographic and biochemical parameters in comparison to the use of open flap debridement alone.

DETAILED DESCRIPTION:
The present study aimed to evaluate the effects of enamel matrix derivatives (EMD) either alone or combined with autogenous bone graft (ABG) applied to intrabony defects in chronic periodontitis patients on clinical/radiographic parameters and gingival crevicular fluid (GCF) transforming growth factor-β1 (TGF-β1) level and, to compare with open flap debridement (OFD). A total of 30 deep intrabony defects in 12 patients were randomly treated with EMD+ABG (Combination group), EMD alone (EMD group) or OFD (Control group). Clinical parameters including plaque index, gingival index, bleeding on probing, probing depth, relative attachment level and recession were recorded at baseline and 6 months post-surgery. Intrabony defect fill percentage was calculated on the standardized radiographs. TGF-β1 level was evaluated in GCF just before surgery and 7, 14, 30, 90, 180 days after surgery using ELISA.

ELIGIBILITY:
Inclusion Criteria:

(a) no systemic diseases as diabetes mellitus or cardiovascular diseases that contraindicated periodontal surgery and could influence the outcome of the therapy; (b) no smoking (c) no medications affecting periodontal tissues; (d) no pregnancy or lactation; (e) a good level of oral hygiene (plaque index < 1, and full mouth bleeding on probing score <20% after initial periodontal treatment), (f) compliance with the maintenance programme and (g) presence of at least one intra-bony defect with a probing depth ≥6 mm, radiographic depth of the defect ≥3 mm as detected on the radiographs.

Exclusion Criteria:

(a) pregnancy or lactating, (b) required an antibiotic premedication, (c) received antibiotic treatment in the previous 6 months, (d) smokers, (e) whose tooth had inadequate amount of attached keratinized gingiva (<1mm)

Ages: 32 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Attachment Gain | 6 months after surgery

SECONDARY OUTCOMES:
Gingival crevicular fluid TGF-β1 level | 1 week, 2 weeks, 4 weeks, 12 weeks and 72 weeks after surgery

OTHER OUTCOMES:
Plaque index | Baseline and 6 months post-surgery.
Gingival index | Baseline and 6 months post-surgery
Bleeding on probing | Baseline and 6 months post-surgery
Probing depth | Baseline and 6 months post-surgery
Relative attachment level | Baseline and 6 months post-surgery
Recession | Baseline and 6 months post-surgery
Intrabony defect fill percentage | Baseline and 6 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Birkan Ağralı, Dr., Principal Investigator — Marmara University Faculty of Dentistry, Department of Periodontology; Bahar Kuru, Prof. Dr., Study Chair — Marmara University, Faculty of Dentistry, Department of Periodontology; Leyla Kuru, Prof. Dr., Study Director — Marmara University, Faculty of Dentistry, Department of Periodontology
Locations (1):
- Marmara University Faculty of Dentistry, Department of Periodontology, Istanbul, Şişli/Nişantaşı, Turkey (Türkiye)